CLINICAL TRIAL: NCT00318435
Title: Fluency Stent-Graft Versus Luminex Stent for Angioplasty of Recurrent Stenosis of the Cephalic Arch in Autogenous Arteriovenous (AV) Access for Hemodialysis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Shaare Zedek Medical Center, Jerusalem , Israel, Shaare Zedek Medical Center, Jerusalem , Israel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2646
Record Dates: First submitted 2006-04-25; First posted 2006-04-26 (Estimated); Last update posted 2008-08-19 (Estimated); Status verified 2006-04

CONDITIONS: Stenosis
MeSH Terms: conditions — Constriction, Pathologic | interventions — Stents

INTERVENTIONS:
Device: Stent or stent-graft deployment

SUMMARY:
The type of hemodialysis access and preservation of this access greatly influences the quality of life and survival of patients undergoing hemodialysis. The Kidney Disease Outcomes Quality Initiative (K/DOQI) guidelines for vascular access recommend the primary placement of native or autogenous hemodialysis fistulas in preference to polytetrafluoroethylene (PTFE) grafts and central venous catheters because the former form of access has fewer complications and a longer durability. However, autogenous hemodialysis fistulas, like polytetrafluoroethylene grafts, are also subject to dysfunction and eventual failure. Endovascular angioplasty has become an accepted alternative treatment to surgical revision for hemodialysis access-related venous stenoses and occlusions. However, the patency rates in the follow-up period are low because of the high frequency of restenosis due to intimal hyperplasia. Since 1988, noncovered stents have been used to improve fistula patency. In the central veins, bare stents demonstrate better patency rates than percutaneous transluminal angioplasty (PTA) alone. Neointimal hyperplasia is the major reason for restenosis following stent placement. The cephalic vein forms the outflow conduit for radiocephalic and brachiocephalic autogenous fistulas. It has recently been suggested that a focal area of the cephalic vein is prone to developing hemodynamically significant stenosis, in what is now termed the cephalic arch. This is the perpendicular portion of the cephalic vein in the region of the deltopectoral groove before its junction with the axillary vein. To overcome the problem of restenosis due to intimal hyperplasia in the cephalic arch the investigators used the insertion of a stent-graft as an alternative approach. In this study they investigated the use of a PTFE-covered nitinol stent-graft (Fluency, Bard) versus a Luminex (Bard) stent.

ELIGIBILITY:
Inclusion Criteria:

* Patients included in this study would be presented for intervention after observation in the Vascular Access Unit for one of the following:

  * the recurrent cephalic arch stenosis identified on periodic duplex scanning, performed by one of the surgeons from the Vascular Access Unit;
  * reduction of flow rate of more than 20% from baseline access flow rate;
  * dynamic venous pressures exceeded threshold levels three consecutive times; or
  * clinical signs (arm swelling, pulsatile fistula, prolonged bleeding from puncture sites) suggesting fistula dysfunction in a patient with previously treated cephalic arch stenosis.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 2006-05; Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Shemesh, MD, Principal Investigator — Shaare Zedek Medical Center
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel

REFERENCES:
- [Derived] Shemesh D, Goldin I, Zaghal I, Berlowitz D, Raveh D, Olsha O. Angioplasty with stent graft versus bare stent for recurrent cephalic arch stenosis in autogenous arteriovenous access for hemodialysis: a prospective randomized clinical trial. J Vasc Surg. 2008 Dec;48(6):1524-31, 1531.e1-2. doi: 10.1016/j.jvs.2008.07.071. Epub 2008 Oct 1. PMID 18829240